CLINICAL TRIAL: NCT01284920
Title: A Phase I/II, Open-Label, Uncontrolled, Dose-Escalation Study of MDV3100 in Patients With Castration-Resistant Prostate Cancer
Brief Title: A Study of MDV3100 to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy of in Prostate Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9785-CL-0111
Record Dates: First submitted 2011-01-18; First posted 2011-01-27 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer; Prostate Neoplasms; Castration Resistant Prostate Cancer (CRPC)
Keywords: docetaxel; Response Evaluation Criteria in Solid Tumor (RECIST); PSA level; MDV3100
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- dose-escalation cohort-1 (Experimental): MDV3100 low dose arm
  Interventions: Drug: MDV3100
- dose-escalation cohort-2 (Experimental): MDV3100 middle dose arm
  Interventions: Drug: MDV3100
- dose-escalation cohort-3 (Experimental): MDV3100 high dose arm
  Interventions: Drug: MDV3100
- dose-expansion cohort (Experimental): dose expansion with MDV3100 middle dose
  Interventions: Drug: MDV3100

INTERVENTIONS:
Drug: MDV3100 — oral

SUMMARY:
This study is to evaluate safety, tolerability pharmacokinetics and efficacy of MDV3100 after oral administration to patients with castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This is a Phase1/2, open-label, uncontrolled study, involving Dose-Escalation Cohorts, where dose will be escalated to next dose with the safety, tolerability, and PK being evaluated in metastatic castration-resistant prostate cancer (mCRPC) patients and an Expansion Cohort, where the efficacy, safety, and PK of MDV3100 in post-chemo mCRPC patients will be evaluated. After evaluation of the safety and tolerability in Dose-Escalation Cohorts, additional patients are included in Expansion Cohort.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Ongoing androgen deprivation therapy with a GnRH analogue or a bilateral orchiectomy
* Progressive disease after prior androgen deprivation therapy (medical or surgical castration)
* For Expansion Cohort, the patient has no more than two prior chemotherapy regimens with at least one regimen containing docetaxel
* For Expansion Cohort, the patient must have measurable lesions by RECIST

Exclusion Criteria:

* Metastases in the brain
* History of another malignancy except for adenocarcinoma of the prostate within the previous 5 years
* Use of bicalutamide within 6 weeks prior to study
* Radiation therapy within 12 weeks prior to study
* Evidence of serious drug hypersensitivity

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-11-02 (Actual); Primary Completion 2012-07-12 (Actual); Study Completion 2014-07-02 (Actual)

PRIMARY OUTCOMES:
Safety assessed by the vital signs, incidence of adverse events, labo-tests and 12-lead EGC | 3 months during the study
  This measure will be assessed on the dose escalation cohorts.
Tumor response assessed by Response Evaluation Criteria in Solid Tumors (RECIST) | Day 85 and end of long term dosing period
  This measure will be assessed on the dose expansion cohort

SECONDARY OUTCOMES:
Prostate Specific Antigen (PSA) Response | Day 85 and end of long term dosing period
Safety assessed by the vital signs, incidence of adverse events, labo-tests and 12-lead ECG | 3 months during the study
  This measure will be assessed on the dose expansion cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kanto
  - Kyusyu
  - Shikoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Akaza H, Uemura H, Tsukamoto T, Ozono S, Ogawa O, Sakai H, Oya M, Namiki M, Fukasawa S, Yamaguchi A, Uemura H, Ohashi Y, Maeda H, Saito A, Takeda K, Naito S. A multicenter phase I/II study of enzalutamide in Japanese patients with castration-resistant prostate cancer. Int J Clin Oncol. 2016 Aug;21(4):773-782. doi: 10.1007/s10147-016-0952-6. Epub 2016 Jan 21. PMID 26793974
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=110